CLINICAL TRIAL: NCT06916091
Title: A Phase 1, Investigator- and Participant-Blinded, Placebo Controlled, Randomized, Single Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Eloralintide (LY3841136) in Chinese Participants With Obesity or Overweight
Brief Title: A Study of Eloralintide (LY3841136) in Chinese Participants With Obesity or Overweight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27320; J3R-MC-YDAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Eloralintide (Experimental): Eloralintide administered subcutaneously (SC)
  Interventions: Drug: Eloralintide
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eloralintide — Administered subcutaneously (SC)
  Other Names: LY3841136
  Arms: Eloralintide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how well Eloralintide (LY3841136) is tolerated and what side effects may occur in overweight and obese Chinese participants. The study drug will be administered subcutaneously (SC) (under the skin). Blood tests will be performed to check how much Eloralintide gets into the bloodstream and how long it takes the body to eliminate it.

The study will last approximately 10 weeks excluding a screening period.

ELIGIBILITY:
Inclusion Criteria:

* Chinese participants. To qualify as Chinese, all 4 of the participant's biological grandparents must be of exclusive Chinese descent and born in China
* Have had a stable body weight for 3 months prior to screening. Participants with body weight change of less than 5% will be allowed
* Have not modified diet or adopted any nutritional lifestyle modification for 3 months before randomization
* Have clinical laboratory test results within a normal range for the population or investigative site at screening and lead-in, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have a body mass index (BMI) within the range 27 to 40 kilogram per square meter (kg/m²)

Exclusion Criteria:

* Are pregnant, or intend to become pregnant or to breastfeed during the study
* Have known allergies to related compounds of eloralintide
* Have any of the following abnormal blood pressure (BP) and/or pulse rate at screening, constituting a risk when taking the investigational product with minor deviations judged to be acceptable by the investigator:

  * Supine BP > 160/90 millimeter mercury (mmHg)
  * Supine pulse rate < 50 or > 100 beats per minute (bpm)
  * Orthostatic hypotension
* Have significant previous or current history of comorbidities capable of significantly altering the absorption, metabolism, or elimination of drugs
* Regularly use known drugs of abuse and/or show positive findings on drug screening that are not consistent with the medical history or concomitant medication history
* Have donated blood of more than 450 mL within the previous 3 months of study screening, or intend to donate blood during the course of the study
* Have a history of chronic medical conditions involving the heart, liver, or kidneys
* Have a medical history or current evidence of clinically significant cardiac condition

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline to Study Completion (Up to 10 Weeks)
  A summary of TEAEs and SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Eloralintide | Baseline to Study Completion (Up to 10 Weeks)
  PK:Cmax of Eloralintide
PK: Area Under the Concentration Versus Time Curve (AUC) of Eloralintide | Baseline to Study Completion (Up to 10 Weeks)
  PK: AUC of Eloralintide

CONTACTS AND LOCATIONS:
Overall Officials: Contact Lilly at 1-800-LillyRx (1-800-545-5979), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/590709